# Incorporating Cardiovascular Risk Assessment into Adolescent & Young Adult Visits to Improve Cardiovascular Health NCT05384834

Date 11/04/2022

## You Are Being Asked to Be in a Research Study

Concise presentation of key concepts

You are being asked to be in a research study. A research study is designed to answer a scientific question. If you agree to be in the study, you will be one of 60 people who are being studied for this specific aim of the study. A total of 100 people are being studied at Emory, Children's Healthcare of Atlanta (CHOA) and the Grady Health System.

## Why is this study being done?

This study is being done to answer the question: Do adolescent and young adult women think that a mobile application used for heart disease prevention is acceptable? You are being asked to be in this research study because you are 13-21 years old and you are at a visit with your doctor.

## Do you have to be in the study?

It is your decision to be part of this research study. You do not have to be in it. Your choice will not affect your access to medical care. Before you make your decision, you should take time to learn about the study.

## What do I have to do if I choose to participate in this study?

If you are eligible and want to be part of the study, you will participate for about three months (two study visits). The researchers will ask you to do the following: answer questions about your health tell us your thoughts about a mobile application used for heart disease prevention. and return for another study visit to answer more questions about your health. ALL of these procedures will be paid for by the study.

## How is this study going to help you?

If you are in the study, you will be helping the researchers answer the study question.

## What are the risks or discomforts I should know about before making a decision?

The study will take time. All studies have some risks. Some risks are relatively small, like being bored or losing time. Some are more serious – for this study, these include loss of privacy, and breach of confidentiality. A full list of expected risks, their frequency and severity are in the "What are the possible risks and discomforts?" section of this document.

Version Date: 10/28/2022

## **Alternatives to Joining This Study**

Since this is not a treatment study, the alternative is not to participate.



## **Costs**

You WILL NOT have to pay for any of the study procedures. Travel expenses will be reimbursed.

## What Should I Do Next?

Read this form, or have it read to you. Make sure the study doctor or study staff explains the study to you. Ask questions (e.g., about exact time commitment, about unfamiliar words, more details on specific procedures, etc.) Take time to consider this and talk about it with your family and friends.

 Version Date: 10/28/2022

## Emory University, Children's Healthcare of Atlanta at Hughes Spalding Hospital, and Grady Health System Consent to be a Research Subject / HIPAA Authorization

<u>Title</u>: Incorporating Cardiovascular Risk Assessment into Adolescent & Young Adult Visits to Improve Cardiovascular Health

IRB Number: 00001418

Principal Investigator: Holly Gooding, MD, MSc

Funding Source: NIH National Heart, Lung, and Blood Institute

If you are the legal guardian of a child who is being asked to participate, the term "you" used in this consent refers to your child

## Introduction

You are being asked to be in a medical research study. This form is designed to tell you everything you need to think about before you decide to consent (agree) to be in the study or not to be in the study. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the research study. You can skip any questions that you do not wish to answer. The decision to join or not join the research study will not cause you to lose any medical benefits. If you decide not to take part in this study, your doctor will continue to treat you.

Before making your decision:

- Please carefully read this form or have it read to you
- Please ask questions about anything that is not clear

You can take a copy of this consent form, to keep. Feel free to take your time thinking about whether you would like to participate. You may wish to discuss your decision with family or friends. Do not sign this consent form unless you have had a chance to ask questions and get answers that make sense to you. By signing this form, you will not give up any legal rights.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

## **Study Overview?**

The purpose of this study is to learn about what adolescent and young adult women think that a mobile application used for heart disease prevention is acceptable.

## **Procedures**

If you want to be in this study, you will be asked to:

- answer questions about your health
- tell us your thoughts about a mobile application used for heart disease prevention
- return for another study visit to answer more questions about your health and record your height, weight and blood pressure.

 IRB Form 06162020 Version Date: 10/28/2022



## **Risks and Discomforts?**

There may be side effects from the study procedures that are not known at this time. The most common risks and discomforts expected in this study are answering questions about alcohol or tobacco use or your health and learning something new about your health.

Rare but possible risks include losing your personal information, or having your personal information stolen. We will do everything we can to make sure that this is unlikely.

## **Benefits**

This study is not designed to benefit you directly. This study is designed to learn more about what teens think about a mobile application that can be used to prevent heart disease. The study results may be used to help others in the future.

## **Compensation**

You will get \$25 for being in the study, even if you cannot finish. This is to compensate you for your time and effort. You will receive an additional \$10 for completing the baseline survey, and an additional \$25 for completing surveys at the three-month study visit for a total of \$35. All travel expenses will be reimbursed.

## **Other Options Outside this Study**

You do not have to be in this study.

## Confidentiality

Certain offices and people other than the researchers may look at study records. Government agencies and Emory employees overseeing proper study conduct may look at your study records. These offices include [the Office for Human Research Protections, the funder(s), the Emory Institutional Review Board, the Emory Office of Compliance]. Study funders may also look at your study records. Emory will keep any research records we create private to the extent we are required to do so by law. A study number rather than your name will be used on study records wherever possible. Your name and other facts that might point to you will not appear when we present this study or publish its results

## **Certificate of Confidentiality**

There is a Certificate of Confidentiality from the National Institutes of Health for this Study. The Certificate of Confidentiality helps us to keep others from learning that you participated in this study. Emory, Children's Healthcare of Atlanta at Hughes Spalding, and Grady Health System will rely on the Certificate of Confidentiality to refuse to give out study information that identifies you. For example, if Emory, Children's Healthcare of Atlanta at Hughes Spalding, or Grady Health System received a subpoena for study records, it would not give out information that identifies you.

The Certificate of Confidentiality does not stop you or someone else, like a member of your family, from giving out information about your participation in this study. For example, if you let your insurance company know that you are in this study, and you agree to give the insurance company research information, then the investigator cannot use the Certificate to withhold this information. This means you and your family also need to protect your own privacy.

The Certificate does not stop Emory, Children's Healthcare of Atlanta at Hughes Spalding, and Grady Health System from making the following disclosures about you:

- Giving state public health officials information about certain infectious diseases,
- Giving law officials information about abuse of a child, elderly person or disabled person.

 IRB Form 06162020



Giving out information to prevent harm to you or others.

Giving the study sponsor or funders information about the study, including information for an audit or evaluation.

## **Storing and Sharing your Information**

De-identified data from this study (data that has been stripped of all information that can identify you) may be placed into public databases where, in addition to having no direct identifiers, researchers will need to sign data use agreements before accessing the data. We will remove or code any personal information that could identify you before your information is shared. This will ensure that, by current scientific standards and known methods, it is extremely unlikely that anyone would be able to identify you from the information we share. Despite these measures, we cannot guarantee anonymity of your personal data.

Your data from this study may be useful for other research being done by investigators at Emory or elsewhere. To help further science, we may provide your deidentified data and/or specimens to other researchers. If we do, we will not include any information that could identify you. If your data or specimens are labeled with your study ID, we will not allow the other investigators to link that ID to your identifiable information.

We will use your sample and data only for research. We will not sell them. However, the results of this research might someday lead to the development of products (such as a mobile application product) that could be sold by a company. You will not receive money from the sale of any such product.

In general, we will not give you any individual results from the study of the samples you give us. If we find something of urgent medical importance to you, we will inform you, although we expect that this will be a very rare occurrence.

## Costs

There will be no costs to you for participating in this study. Transportation costs will be covered by the study. You will not be charged for any of the research activities.

## Withdrawal from the Study

You have the right to leave a study at any time without penalty.

The researchers also have the right to stop your participation in this study without your consent for any reason, especially if they believe it is in your best interest or if you were to object to any future changes that may be made in the study plan.

 Version Date: 10/28/2022



## Authorization to Use and Disclose Protected Health Information

The privacy of your health information is important to us. As part of this study, we will be requesting health care entities who are covered by the Health Insurance Portability and Accountability Act and regulations (HIPAA) to provide us with health information that identifies you ("individually identifiable health information" or "IIHI"). Because the health care entities are covered by HIPAA, we must have your authorization to obtain your IIHI from them. However, the researchers who get your IIHI from the health care entities are not covered by HIPAA. Once they receive your IIHI from the health care entities, they will put it in a separate research record that is not a part of your medical record. IIHI placed in the separate research record is not be covered by HIPAA.

## **Purpose of this Authorization:**

By signing this form, you give us permission to get your IIHI from health care entities and to use and share your IIHI as described in this document. You do not have to sign this form. If you do not sign this form, then you may not participate in the research study.

## **No Provision of Treatment**

There is no research-related treatment involved in this study. You may receive any non-research related treatment whether or not you sign this form.

## IIHI that Will be Used/Disclosed:

The IIHI that we will use or share for the research study includes:

- Medical information about you including your medical history
- Date of doctor's visits

## Purposes for Which Your IIHI Will be Used/Disclosed:

We will use and share your IIHI for the conduct and oversight of the research study. Once we have your IIHI we will keep it in a separate research record that will be used for the conduct of the study. If you leave the study, we may use your IIHI to determine your vital status or contact information.

## Use and Disclosure of Your IIHI That is Required by Law:

We will use and disclose your IIHI when we are required to do so by law. This includes laws that require us to report child abuse or abuse of elderly or disabled adults. We will also comply with legal requests or orders that require us to disclose your IIHI. These include subpoenas or court orders.

## People Who will Use/Disclose Your IIHI:

The following people and groups will use and disclose your IIHI in connection with the research study:

- The Principal Investigator and the research staff will use and disclose your IIHI to conduct the study.
- Emory may use and disclose your IIHI to get payment for conducting the study and to run normal business operations.
- The Principal Investigator and research staff will share your IIHI with other people and groups to help
  conduct the study or to provide oversight for the study. This includes sharing your IIHI with people and
  groups at other sites who are helping conduct the study.

 IRB Form 06162020



- The NIH National Heart, Lung, and Blood Institute is the Sponsor of the study. The Sponsor may use and disclose your IIHI to make sure the research is done correctly and to collect and analyze the results of the research. The Sponsor may disclose your IIHI to other people and groups like study monitors to help conduct the study or to provide oversight for the study.
- The following people and groups will use your IIHI to make sure the research is done correctly and safely:
  - Emory, Grady Health System, and Children's Healthcare of Atlanta offices that are part of the Human Research Participant Protection Program and those that are involved in study administration. These include the Emory and Children's Healthcare of Atlanta IRB, the Emory University and Healthcare Compliance Offices, the Grady Research Oversight Committee, the Emory Office for Clinical Research.
  - o Government agencies that regulate the research including: Office for Human Research Protections.
  - Public health agencies.
  - Research monitors and reviewer.
  - Accreditation agencies.
- Sometimes a Principal Investigator or other researcher moves to a different institution. If this happens, your IIHI may be shared with that new institution and their oversight offices.

## **Expiration of Your Authorization**

Your IIHI will be used until this research study ends.

## **Revoking Your Authorization**

If you sign this form, at any time later you may revoke (take back) your permission to use your IIHI. If you want to do this, you must contact the study team at:

At that point, the researchers would not collect any more of your IIHI. But they may use or disclose the information you already gave them as described in this Authorization. If you revoke your authorization you will not be able to stay in the study.

## Other Items You Should Know about Your Privacy

Not all people and entities are covered by the Privacy Rules. HIPAA only applies to health care providers, health care payers, and health care clearinghouses. HIPAA does not apply to research that does not include treatment that is billed to insurers or government benefit programs. If we disclose your information to people who are not covered by the Privacy Rules, including HIPAA, then your information won't be protected by the Privacy Rules. People who do not have to follow the Privacy rules can use or disclose your information with others without your permission if they are allowed to do so by the laws that cover them. The researchers, the Sponsor, and people and companies working with them are not covered by the Privacy Rules. They will only use and disclose your information as described in this Consent and Authorization.

To maintain the integrity of this research study, you generally will not have access to your IIHI related to this research until the study is complete. When the study ends, and at your request, you generally will only have access to your IIHI that we maintain in a designated record set. A designated record set is data that includes medical information or billing records that your health care providers use to make decisions about you. You will not have a right of access to IIHI kept in a separate research record used only for research purposed. If it is necessary for your health care, your health information will be provided to your doctor.

 We may remove identifying information from your IIHI. Information without identifiers is not subject to HIPAA and may be used or disclosed with other people or organizations for purposes besides this study.

 Version Date: 10/28/2022



## **Contact Information**

Contact Dr. Holly Gooding at

- if you have any questions about this study or your part in it,
- if you have questions, concerns or complaints about the research

Contact the Emory Institutional Review Board at

- if you have questions about your rights as a research participant.
- if you have questions, concerns or complaints about the research.

You may also let the IRB know about your experience as a research participant through our Research Participant Survey at <a href="https://tinyurl.com/ycewgkke">https://tinyurl.com/ycewgkke</a>.

If you are patient receiving care from the Grady Health System and you have a question about your rights, you may contact the Office of Research Administration at research@gmh.edu.

# TO BE FILLED OUT BY SUBJECT ONLY Please print your name, sign, and date below if you agree to be in this research study. By signing this consent and authorization form, you will not give up any of your legal rights. We will give you a copy of the form to keep. Name of Subject Signature of Subject (18 or older and able to consent) Date Time Signature of Legally Authorized Representative Date Time Authority of Legally Authorized Representative or Relationship to Subject TO BE FILLED OUT BY STUDY TEAM ONLY Name of Person Conducting Informed Consent Discussion

 Version Date: 10/28/2022

Date

Time

**Signature of Person Conducting Informed Consent Discussion** 



 Version Date: 10/28/2022 IRB Form 06162020